CLINICAL TRIAL: NCT07291518
Title: Influence of Menstrual Cycle Phases on Post-Endodontic Pain: A Comparative Clinical Study With Male Patients
Brief Title: Post-Endodontic Pain According to Menstrual Cycle Phases
Acronym: PEP-MC
Status: Completed | Type: Observational
Sponsor: Ahter Sanal Cikman (Other)
Responsible Party: Sponsor-Investigator, Ahter Sanal Cikman, Principal Investigator (PI), Assistant Professor of Endodontics, Recep Tayyip Erdogan University
Organization: Recep Tayyip Erdogan University (Other)
Other Study IDs: MCOBAN-ENDO2025; 2023/184 (Ethics Approval) (Other: Recep Tayyip Erdogan University Ethics Committee)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Root Canal Treatment
Keywords: Endodontic treatment; Post-endodontic pain; Pain perception; Mandibular molars; Dental pain; postoperative pain; Menstrual cycle
MeSH Terms: conditions — Toothache; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: root canal treathment — All participants underwent standard root canal treatment under local anesthesia and rubber dam isolation. Root canals were prepared using ProTaper Next rotary files, irrigated with 2.5% sodium hypochlorite and 17% EDTA, dried with paper points, and filled using a sealant and gutta-percha. The teeth were then restored coronally with composite resin. Postoperative pain and analgesic use were monitored for 72 hours to assess the influence of menstrual cycle phase on pain perception. This standardized procedure ensures consistency across participants and allows comparisons between menstrual phases and between male patients.

SUMMARY:
This study aimed to evaluate whether the phase of the menstrual cycle affects pain after root canal treatment. A total of 99 patients (72 females and 27 males) who needed root canal treatment in lower molar teeth were included. Female participants were grouped according to their menstrual cycle phase: menstrual, proliferative, and secretory. All patients received the same endodontic treatment procedure under local anesthesia. Postoperative pain intensity was recorded using a Visual Analog Scale (VAS) at 8 hours, 8-24 hours, 24-48 hours, and 48-72 hours after treatment. Analgesic (ibuprofen) use was also recorded. The results showed that women in the menstrual and secretory phases experienced higher pain levels than men, while pain levels in the proliferative phase were similar to those in men. The findings suggest that the menstrual cycle phase may influence short-term pain perception after root canal treatment.

DETAILED DESCRIPTION:
This prospective clinical study investigates the effect of menstrual cycle phase on postendodontic pain intensity in female patients compared to male patients. Ninety-nine participants requiring endodontic treatment for asymptomatic necrotic mandibular molars were enrolled in the study. Female participants were categorized into menstrual, proliferative, or secretory phases based on the first day of their last menstrual period. All treatments were standardized and performed under local anesthesia with rubber dam isolation, including root canal preparation using rotary files, irrigation with 2.5% sodium hypochlorite and 17% EDTA, and obturation with root canal sealer. Postoperative pain was self-assessed using a Visual Analog Scale (VAS) at multiple time points for up to 72 hours, and analgesic consumption was recorded. Data were analyzed with nonparametric tests to compare pain levels across cycle phases and in male participants. This study provides detailed information on potential hormonal influences on postoperative pain and may guide clinicians in planning endodontic treatments to maximize postoperative comfort in female patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Male or female patients requiring endodontic treatment of asymptomatic
* Necrotic mandibular first or second molars
* Female patients with regular menstrual cycles
* Patients who have not taken analgesics in the last 3 days
* Patients willing to provide written informed consent

Exclusion Criteria:

* Smoking habit
* Systemic diseases or use of systemic drugs
* Parafunctional habits such as bruxism
* Preoperative pain
* Teeth requiring prosthetic restoration
* Teeth with external or internal resorption
* Immature teeth
* Periodontal probing depth > 3 mm
* Pregnant women
* Women with irregular menstrual cycles
* Patients who refuse to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study population consists of 99 adult patients (72 females and 27 males), aged 18-50 years, requiring endodontic treatment for asymptomatic necrotic mandibular first or second molars. Female participants have regular menstrual cycles and are categorized into menstrual, proliferative, or secretory phases. Patients with systemic diseases, smoking habits, preoperative pain, parafunctional habits, teeth requiring prosthetic restoration, immature teeth, periodontal probing depth greater than 3 mm, or irregular menstrual cycles are excluded. All participants provided written informed consent prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Post-Endodontic Pain Intensity | Up to 72 hours post-treatment.
  Measured using Visual Analog Scale (VAS) at 8 hours, 8-24 hours, 24-48 hours, and 48-72 hours after root canal treatment. Participants self-recorded the highest pain intensity at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Çoban Öksüzer, Principal Investigator — pamukkale univercity; Ömer Hatipoğlu, Study Director — recep tayyip erdoğan univercity; Fatma Pertek Hatipoğlu, Study Director — recep tayyip erdoğan univercity; ahter şanal çıkman, Study Director — recep tayyip erdoğan univercity
Locations (1):
- Recep Tayyip Erdoğan Univercity, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.aae.org/patients/root-canal-treatment/